CLINICAL TRIAL: NCT06641427
Title: Different Aspects and Etiologies of Gastointestinal Bleeding in Patients With Systemic Lupus Erythematosus
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mina Noshy Baskales, Dr, Assiut University
Other Study IDs: GIT bleeding in SLE patients
Record Dates: First submitted 2024-10-12; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The association between SLE and development of of gastrointestinal bleeding

DETAILED DESCRIPTION:
systemic lupus erythematosus (SLE) is an autoimmune disease characterized by multisystem inflammation, variable clinical manifestations, and a variable clinical course. It affects multiple systems and can occasionally manifest as hematological disorders and gastrointestinal (GI) tract abnormalities(1). The complications of SLE are diverse and severe, and may include lupus pneumonitis, lupus encephalopathy, intestinal pseudo-obstruction, gastrointestinal bleeding, and vasculitis (2) . The potential severity of SLE-related GI manifestations is concerning, considering that more than 50% of SLE patients develop GI symptoms at some point during the course of illness. The incidence and prevalence of GI involvement during the course of SLE disease vary widely. This could be due to less attention being paid to GI manifestations than other organ symptoms, such as lupus nephritis. According to an autopsy study, 60-70% of SLE patients had evidence of peritonitis, whereas only 10% showed clinical manifestations throughout their lives(3). Any part of the GI tract and the hepatobiliary system can be involved from the mouth to the anus. The liver can also be affected by SLE; abnormal liver function test results were obtained in 23%-79% of cases and hepatomegaly in 39%-40%. In terms of risk factors for GI involvement in SLE, SLE patients with Raynaud's phenomenon, hypocomplementemia, and positive anti-neutrophil cytoplasmic antibody were at increased risk of developing GI complications(4). The main pathological mechanisms of GI involvement in SLE involved mesenteric vasculitis, intestinal pseudo-obstruction and protein losing enteropathy(5). There is a wide variation of GI manifestations, including gastro-esophageal reflux, dysphagia, abdominal pain, constipation, diarrhea, faecal incontinence, intestinal pseudo-obstruction (IPO), perforations, and haemorrhage. When GI presents as the initial affected system of SLE, there is likely to be a delay in the diagnosis(6). Clinical presentations of GI lupus are non-specific and can be difficult to differentiate from infective, thrombotic, therapy-related and non-SLE aetiologies(7).

ELIGIBILITY:
Inclusion Criteria:

- Patient more than 18 years old classified as systemic lupus erythematosus Both sex

Exclusion Criteria:

* Patients with other clinical conditions that causes gastrointestinal bleeding as ulcerative colitis & chrons

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient more than 18 years old classified as systemic lupus erythematosus Both sex with no other clinical conditions that causes gastrointestinal bleeding as ulcerative colitis & chrons
Sampling Method: Non-Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
review diferrent aspects and causes of GIT bleeding in SLE patient | baseline
  in this study we will review diferrent aspects and causes of GIT bleeding in SLE patient

CONTACTS AND LOCATIONS:
Overall Officials: Zine alabden Ahmed Said, Principal Investigator — Assiut University; Eman Mohamed Ebrahem, Principal Investigator — Assiut University